CLINICAL TRIAL: NCT07201584
Title: A Comparative Bioavailability of Two Torasemide 10 mg Tablets Formulations in Healthy Adult Participants Under Fasting Conditions: a Prospective, Open-label, Randomized, Single-dose, Two-treatment, Two-period, Two-sequence, Crossover Bioequivalence Study
Brief Title: A Comparative Bioavailability Study of Two Torasemide 10 mg Tablets Formulations in Healthy Adult Participants Under Fasting Conditions:
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Berlin-Chemie AG Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BCKZ/24/Tor-BE/001
Record Dates: First submitted 2025-09-10; First posted 2025-10-01 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Male and Female Volunteers
Keywords: Torasemide; Bioequivalence
MeSH Terms: interventions — Torsemide

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, open-lable, , single-dose, two-period, two-treatment, two-sequence, crossover bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Torasemide 10 mg tablet (Experimental): Single dose administration (10 mg) with 240 mL of water under fasting conditions
  Interventions: Drug: Torasemide tablet 10 mg
- Unat® 10 (Torasemide) tablets (Viatris Healthcare GmbH) (Experimental): Single dose administration (10 mg) with 240 mL of water under fasting conditions
  Interventions: Drug: Unat® 10 tablets (Torasemide 10 mg)

INTERVENTIONS:
Drug: Torasemide tablet 10 mg — Tablets by Berlin-Chemie AG (Germany)
  Arms: Torasemide 10 mg tablet
Drug: Unat® 10 tablets (Torasemide 10 mg) — Tablets by Viatris Healthcare GmbH (Germany)
  Arms: Unat® 10 (Torasemide) tablets (Viatris Healthcare GmbH)

SUMMARY:
The purpose of this study is to evaluate the bioavailability, safety and tolerability of Torasemide 10 mg tablets (Berlin-Chemie AG), compared to Unat® 10 tablets (Viatris Healthcare GmbH) in healthy adult participants under fasting conditions.

DETAILED DESCRIPTION:
In this Phase I study, the test medication Torasemide 10 mg tablets (Berlin-Chemie AG) is compared to Unat® 10 tablets (Viatris Healthcare GmbH) in terms of bioequivalence of the tested formulations under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female individuals aged 18 to 55 years inclusive at the time of signing the ICF.
2. Body weight ≥50 kg and Body Mass Index (BMI) between ≥18.5 and <30.0 kg/m2.
3. A healthy individual as determined by the Investigator based on medical history and results of standard clinical, laboratory and instrumental methods of examination (individuals with not clinically significant [NCS] abnormalities are eligible for the study).
4. A non-smoker (for at least 3 months before screening), verified by the cotinine test at screening.
5. A negative urine pregnancy test (rapid test) within 24 h before the first IMP dose for female individuals of childbearing potential. Postmenopausal (no menses for at least 1 year) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) females are exempted from the requirement.
6. Individuals with preserved reproductive potential should agree to use, with their partner, adequate contraception throughout the study and for 30 days thereafter (contraceptive methods with reliability greater than 90%: cervical caps with spermicide, diaphragms with spermicide, condoms with intravaginal spermicide, non-hormonal intrauterine devices), or true sexual abstinence.
7. Capable of understanding the ICF and giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and the study protocol.

Exclusion Criteria:

1. Known hypersensitivity or intolerance to torasemide, other sulfonylureas, or any other excipient of the IMPs.
2. History of renal failure with anuria.
3. History of hepatic precoma, coma.
4. History of hypotension.
5. History of hypovolemia.
6. History of hyponatremia and/or hypokalemia.
7. History of substantial micturition disorders (e.g. due to prostatic hypertrophy).
8. History of gout.
9. History of cardiac arrhythmias (e.g. SA block, 2nd or 3rd degree AV block).
10. History of latent or manifest diabetes mellitus or any form of hyperglycemia.
11. History of pathological changes in the acid-base balance.
12. History of pathological changes in the blood count (e.g. thrombocytopenia, anemia in patients without renal insufficiency).
13. History of abnormally high (≥190 mg/dL [≥4.9 mmol/L]) low-density lipoprotein (LDL) cholesterol levels within 3 months before the first IMP dose.
14. Abnormally high triglycerides levels (>150 mg/dL [>1.7 mmol/L]) within 3 months before the first IMP dose.
15. History of renal insufficiency (creatinine clearance between 20 mL and 30 mL/min and/or serum creatinine concentrations between 3.5 mg/dL and 6 mg/dL) due to nephrotoxic substances.
16. History of other clinically significant cardiovascular, respiratory, renal, hepatic, endocrine, metabolic, gastrointestinal, hematological, genito-urinary disease, bleeding disorders, neurological or psychiatric pathology, oncologic disease, autoimmune disease, dermatological disease or other chronic disease, that makes the individual ineligible for the study.
17. Acute infectious diseases (e.g. influenza, acute respiratory bacterial or viral infections incl. COVID-19) less than 4 weeks before the first IMP dose.
18. Hereditary galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.
19. Systolic blood pressure < 90 mmHg or ≥ 130 mmHg and/or diastolic blood pressure < 60 mmHg or ≥ 85 mmHg.
20. Heart rate < 60 or > 100 beats per minute.
21. The presence of any other condition which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
22. Use of the following medications within the relevant period before the first IMP dose:

    1. Use of medications (including hormonal contraceptives) that have a significant effect on circulatory dynamics, liver function, etc. (barbiturates, omeprazole, cimetidine, non-steroidal anti-inflammatory drugs, angiotensin-converting enzyme inhibitors, angiotensin II receptor antagonists, diuretics, etc.) within 2 months before the first IMP dose.
    2. Use of depot-forms of any medications within 3 months before the first IMP dose.
    3. Use of any other prescribed or non-prescribed medication, herbal remedies, vitamins and minerals within 2 weeks before the first IMP dose or longer (at least 5 elimination half-lives) if the medication has a long half-life.
23. Female individuals who are lactating.
24. Female individuals of childbearing potential, having unprotected sexual intercourse with any unsterilized male partner (i.e., a man who is not sterilized by vasectomy for at least 6 months) within 30 days before the first IMP dose.
25. Blood donation/blood loss >450 mL within 60 days or apheresis donation within 30 days before the first IMP dose.
26. Dehydration (e.g. due to diarrhea, vomiting, or other causes) within the last 48 h before the first IMP dose.
27. Positive test result for COVID-19 rapid antigen test at admission to the Study Site.
28. Positive test results for HIV or hepatitis B (HBsAg, anti-HBc) or C (anti-HCV) or syphilis at screening.
29. History of drug or alcohol abuse within 1 year before the screening. Alcohol abuse is defined as regular intake of more than 10 units of alcohol a week (1 unit equivalent to 200 mL of dry wine or 50 mL of strong alcoholic drinks or 500 mL of beer).
30. Positive screen for drugs or alcohol at screening.
31. Individuals who have been on a special diet (for whatever reason, e.g. vegetarians or hypocaloric diet [< 1000 kcal/day]) within the 28 days before the first IMP dose and throughout the study.
32. Intake of methylxanthine-containing substances (e.g., coffee, tea, chocolate, cocoa, energy drinks, cola) as well as citrus fruits and cranberry (including juices, fruit drinks, etc.) within the last 48 h before the first IMP dose.
33. Intake of food or beverages containing poppy seeds within 72 h before the first IMP dose.
34. Excessive consumption (defined as greater than 6 servings - 1 serving being approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks or other caffeinated beverages per day within 2 weeks before the first IMP dose.
35. Mental, physical and other reasons that do not allow the individual, according to Investigator's opinion, to assess their behavior adequately, to follow correctly the requirements of the clinical study protocol and to assess the expected risks and possible discomfort.
36. Participation in another clinical study (except if no investigational product was administered) within 3 months before the first IMP dose.
37. Employee or family member of the Sponsor or the involved Contract Research Organization (CRO) or the Study Site.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
C max | 24 hours
  Maximum plasma concentration
AUC 0-last | 24 hours
  Area under the curve from time 0 to the last quantifiable time point

SECONDARY OUTCOMES:
AUC 0-Inf | Through study completion, an average of 1 year
  Area under the curve from time 0 to infinity
T max | 24 hours
  Time to maximum plasma concentration
C last | 24 hours
  Last observed quantifiable concentration
T last | 24 hours
  Time to last quantifiable concentration
T lag | 24 hours
  Lag time
λz | 24 hours
  Terminal elimination rate constant
T 1/2 | 24 hours
  Elimination half-life
Residual area | 24 hours
  Residual area under the plasma concentration curve

OTHER OUTCOMES:
Analysis of Adverse Events (AEs) | 28 days
  Number (%) of subjects with Adverse Events
Analysis of Adverse Events (AEs) | 28 days
  Number (%) of subjects with drug-related AEs
Analysis of Adverse Events (AEs) | 28 days
  Number (%) of subjects withrawn from the study due to drug-related AEs
Analysis of Adverse Events (AEs) | 28 days
  Number (%) of subjects with Serious Adverse Events (SAEs)
Analysis of Adverse Events (AEs) | 28 days
  Number (%) of subjects withdrawn due to drug-related Serious Adverse Events (SAEs)
Analysis of Adverse Events (AEs) | 28 days
  Number (%) of subjects withrawn from the study due to AEs

CONTACTS AND LOCATIONS:
Overall Officials: Guldana Abdullaeva, MD, Principal Investigator — LLP MedStartUp, Ili district, Otegen Batyr settlement, Industrial Zone 200A, Almaty region
Locations (1):
- LLP MedStartUp, Almaty, Ili District, Otegen Batyr Settlement, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
No publication in an ICMJE journal is planned

REFERENCES:
- See also: Related Info — https://www.menarini.com/en-us/innovation-research/clinical-trials/clinical-trials-database.html